CLINICAL TRIAL: NCT00244309
Title: A Randomized Trial of Tamsulosin and/or Dutasteride Versus Placebo to Relieve Urinary Symptoms After Brachytherapy for the Treatment of Localized Prostate Cancer
Brief Title: Study of Tamsulosin and/or Dutasteride to Relieve Urinary Symptoms After Brachytherapy for Localized Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Jay Ciezki, Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CASE14804; GSK106046 (formerly 103988)
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
Keywords: brachytherapy; urinary symptoms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tamsulosin and/or dutasteride

SUMMARY:
The purpose of this study is to determine whether a drug named tamsulosin (Flomax), or another drug named dutasteride (Avodart), or a combination of these two drugs is effective in improving urinary symptoms and decreasing the rate of intermittent self-catheterization after prostate brachytherapy.

DETAILED DESCRIPTION:
Image-guided transperineal permanent prostate brachytherapy (PI) is an accepted curative treatment option for patients with early stage prostate cancer. The most severe side effect of PI is urinary retention requiring intermittent self-catheterization (ISC). This study will assess the ability of pharmacologic intervention to ameliorate the post-operative side effect of PI. The use of both tamsulosin and dutasteride is proposed to have benefit in reducing urinary symptom score and in reducing the rate of intermittent self-catheterization for patients with prostate adenocarcinoma after prostate implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible for a prostate implant
* Patient is greater than 18 years of age
* Patient is able to give informed consent
* Patient does not currently take Flomax, Dutasteride or Finasteride
* Patient does not have a known hypersensitivity reaction to Flomax or Dutasteride

Exclusion Criteria:

* Patients who have a known hypersensitivity reaction to tamsulosin, dutasteride or finasteride and those patients who are already on any prior to prostate implantation
* Patients who are taking a PDE-5 inhibitor including sildenafil (Viagra), tadalafil (Cialis) and vardenafil (Levitra) are ineligible to participate unless they are willing to discontinue using those drugs one week prior to their implant and for three months after the implant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
AUA score will be used to assess severity of urinary symptoms. All patients will be contacted weekly by telephone for 12 weeks then monthly postoperatively to get their AUA score. A total of 21 AUA scores postoperatively.

SECONDARY OUTCOMES:
Use of intermittent self-catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Jay P Ciezki, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ragde H, Blasko JC, Grimm PD, Kenny GM, Sylvester JE, Hoak DC, Landin K, Cavanagh W. Interstitial iodine-125 radiation without adjuvant therapy in the treatment of clinically localized prostate carcinoma. Cancer. 1997 Aug 1;80(3):442-53. doi: 10.1002/(sici)1097-0142(19970801)80:33.0.co;2-x. PMID 9241078
- [Background] Ragde H, Korb LJ, Elgamal AA, Grado GL, Nadir BS. Modern prostate brachytherapy. Prostate specific antigen results in 219 patients with up to 12 years of observed follow-up. Cancer. 2000 Jul 1;89(1):135-41. PMID 10897010
- [Background] Blasko JC, Ragde H, Grimm PD. Transperineal ultrasound-guided implantation of the prostate: morbidity and complications. Scand J Urol Nephrol Suppl. 1991;137:113-8. PMID 1947828
- [Background] Kleinberg L, Wallner K, Roy J, Zelefsky M, Arterbery VE, Fuks Z, Harrison L. Treatment-related symptoms during the first year following transperineal 125I prostate implantation. Int J Radiat Oncol Biol Phys. 1994 Mar 1;28(4):985-90. doi: 10.1016/0360-3016(94)90119-8. PMID 8138452
- [Background] Terk MD, Stock RG, Stone NN. Identification of patients at increased risk for prolonged urinary retention following radioactive seed implantation of the prostate. J Urol. 1998 Oct;160(4):1379-82. PMID 9751358
- [Background] Benoit RM, Naslund MJ, Cohen JK. A comparison of complications between ultrasound-guided prostate brachytherapy and open prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):909-13. doi: 10.1016/s0360-3016(00)00506-x. PMID 10863059
- [Background] Lee N, Wuu CS, Brody R, Laguna JL, Katz AE, Bagiella E, Ennis RD. Factors predicting for postimplantation urinary retention after permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1457-60. doi: 10.1016/s0360-3016(00)00784-7. PMID 11121648
- [Background] Bruno JF, Whittaker J, Song JF, Berelowitz M. Molecular cloning and sequencing of a cDNA encoding a human alpha 1A adrenergic receptor. Biochem Biophys Res Commun. 1991 Sep 30;179(3):1485-90. doi: 10.1016/0006-291x(91)91740-4. PMID 1656955
- [Background] Ramarao CS, Denker JM, Perez DM, Gaivin RJ, Riek RP, Graham RM. Genomic organization and expression of the human alpha 1B-adrenergic receptor. J Biol Chem. 1992 Oct 25;267(30):21936-45. PMID 1328250
- [Background] Lepor H. Phase III multicenter placebo-controlled study of tamsulosin in benign prostatic hyperplasia. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):892-900. doi: 10.1016/s0090-4295(98)00126-5. PMID 9609623
- [Background] Lepor H. Long-term evaluation of tamsulosin in benign prostatic hyperplasia: placebo-controlled, double-blind extension of phase III trial. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):901-6. doi: 10.1016/s0090-4295(98)00127-7. PMID 9609624
- [Background] Chapple CR, Wyndaele JJ, Nordling J, Boeminghaus F, Ypma AF, Abrams P. Tamsulosin, the first prostate-selective alpha 1A-adrenoceptor antagonist. A meta-analysis of two randomized, placebo-controlled, multicentre studies in patients with benign prostatic obstruction (symptomatic BPH). European Tamsulosin Study Group. Eur Urol. 1996;29(2):155-67. PMID 8647141
- [Background] Schulman CC, Cortvriend J, Jonas U, Lock TM, Vaage S, Speakman MJ. Tamsulosin, the first prostate-selective alpha 1A-adrenoceptor antagonist. Analysis of a multinational, multicentre, open-label study assessing the long-term efficacy and safety in patients with benign prostatic obstruction (symptomatic BPH). European Tamsulosin Study Group. Eur Urol. 1996;29(2):145-54. PMID 8647140
- [Background] Prosnitz RG, Schneider L, Manola J, Rocha S, Loffredo M, Lopes L, D'Amico AV. Tamsulosin palliates radiation-induced urethritis in patients with prostate cancer: results of a pilot study. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):563-6. doi: 10.1016/s0360-3016(99)00246-1. PMID 10524406
- [Background] Elshaikh MA, Angermeier K, Ulchaker JC, Klein EA, Chidel MA, Mahoney S, Wilkinson DA, Reddy CA, Ciezki JP. Effect of anatomic, procedural, and dosimetric variables on urinary retention after permanent iodine-125 prostate brachytherapy. Urology. 2003 Jan;61(1):152-5. doi: 10.1016/s0090-4295(02)02142-8. PMID 12559287
- [Background] Nag S, Beyer D, Friedland J, Grimm P, Nath R. American Brachytherapy Society (ABS) recommendations for transperineal permanent brachytherapy of prostate cancer. Int J Radiat Oncol Biol Phys. 1999 Jul 1;44(4):789-99. doi: 10.1016/s0360-3016(99)00069-3. PMID 10386635
- [Background] Nag S, Bice W, DeWyngaert K, Prestidge B, Stock R, Yu Y. The American Brachytherapy Society recommendations for permanent prostate brachytherapy postimplant dosimetric analysis. Int J Radiat Oncol Biol Phys. 2000 Jan 1;46(1):221-30. doi: 10.1016/s0360-3016(99)00351-x. PMID 10656396